CLINICAL TRIAL: NCT03547570
Title: Progressive Heavy Shoulder Resistance Training for Patients With Hypermobility Spectrum Disorders and Shoulder Symptoms: a Feasibility Study
Brief Title: Resistance Training for Patients With Hypermobility Spectrum Disorders and Shoulder Symptoms: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Esbjerg Municipality (Other Government); Region of Southern Denmark (Other); The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Behnam Liaghat, Principal Investigator, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20170066
Record Dates: First submitted 2018-05-03; First posted 2018-06-06 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Hypermobility Syndrome Shoulder; Shoulder Pain Chronic
Keywords: Joint instability; Hypermobility; Shoulder; Strength training
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Intervention Model Description: Intervention group only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heavy shoulder resistance training (Experimental): Progressive heavy shoulder resistance training performed twice a week at the physiotherapy clinic under supervision, while once weekly training at home will be recommended.
  Interventions: Other: Progressive heavy shoulder resistance training

INTERVENTIONS:
Other: Progressive heavy shoulder resistance training — The training programme includes five exercises identified in literature to target scapular and rotator cuff muscles.

SUMMARY:
Hypermobility Spectrum Disorders (HSD) is a recent diagnosis that covers joint hypermobility with one or more secondary symptomatic musculoskeletal manifestations. Current clinical management of this population with shoulder symptoms is a non-standardized combination of physiotherapy modalities including exercise prescription. There is evidence suggesting that progressive heavy resistance training increases muscle strength and tendon stiffness, which may be valuable for treatment of this population.

The aim of this study is to evaluate the feasibility of progressive heavy shoulder resistance training (PHSRT) for adults with HSD and shoulder symptoms.

DETAILED DESCRIPTION:
Hypermobility Spectrum Disorders (HSD) is a recent diagnosis that covers joint hypermobility with one or more secondary symptomatic musculoskeletal manifestations. Current clinical management of this population with shoulder symptoms is a non-standardized combination of physiotherapy modalities including exercise prescription. There is evidence suggesting that progressive heavy resistance training increases muscle strength and tendon stiffness, which may be valuable for treatment of this population.

The aim of this study is to evaluate the feasibility of progressive heavy shoulder resistance training (PHSRT) for adults with HSD and shoulder symptoms before safely performing a definitive RCT-study in a large cohort. The objectives are to address whether PHSRT is feasible regarding i) patient recruitment and retention, ii) adherence to exercise protocol and its progression levels, iii) completion of objective outcome measures, and iv) registering potential flare up in shoulder symptoms.

Study progression criteria are based on a traffic light system of green (go), amber (amend) and red (stop). Results of these progression criteria will be evaluated by the investigator group, who will recommend amendments that need to be made before proceeding with the definitive RCT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 65
* Generalized HSD (G-HSD) defined with Beighton score cut-off ≥ 5 for women up to the age of 50 years and ≥ 4 for those above 50 years and all men [21, 22] or historical HSD (H-HSD) if the Beighton score was 1 point below the age and sex-specific cut-off AND the five-part questionnaire (5PQ) was positive (= at least two positive items). In patients with acquired joint limitations (past surgery, wheelchair, amputations) affecting the Beighton score calculation, the assessment of GJH only included a positive 5 part-questionnaire.
* Present with one or more secondary symptomatic musculoskeletal manifestations, defined as either musculoskeletal pain in minimum one shoulder for at least three months or recurrent joint dislocations or joint instability without a reported history of trauma defined as: a) minimum three atraumatic dislocations in same shoulder or minimum two atraumatic dislocations in two different joints (minimum one in the shoulder) occurring at different times, or b) medical confirmation of joint instability in minimum two joints (minimum one in the shoulder) not related to trauma.

Exclusion Criteria:

* Clinically suspected referred pain from the cervical spine
* Systemic rheumatic diseases (e.g. Marfans, Stickler's or Loeys Dietz syndromes)
* Neurological diseases
* Pregnancy or childbirth within the latest year
* Shoulder surgery within the past year
* Inability to speak and understand Danish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Patient recruitment | 4 months
  Green: Inclusion rate of one patient per general practitioner or physiotherapist every month (approximately n=6-8/month).
  Amber: If the recruitment rate falls behind, screening logs and reasons for exclusion will be explored after the first month in order to adjust eligibility criteria (n<6 after first month)
  Red: No recruitment after two months
Completion of the outcome measures | Baseline measures
  Green: 120 minutes for completing all objective outcome measures and at least 67% of patients answering that it was an acceptable duration
  Amber: Between 121-150 minutes or between 50-66% of patients answering that it was an acceptable duration
  Red: >150 minutes or <50% of patients answering that it was an acceptable duration
Patient retention | 4 months
  Green: 10 or more patients show up at 16-weeks follow up
  Amber: 6-9 patients show up at 16-weeks follow up
  Red: Less than 6 patients show up at 16-weeks follow up
Adherence to training intervention | 4 months
  Green: At least 75% of patients adhering to at least 75% of training sessions
  Amber: 50-75% of patients adhering to 50-75% of training sessions
  Red: <50% of patients adhering to <50% of training sessions
Adverse events | 4 months
  Green: No or minor adverse events with no patients discontinuing the trial
  Amber: Minor or serious adverse events leading to 2 or less patients discontinuing the trial
  Red: Serious adverse events leading to >2 patients discontinuing the trial

SECONDARY OUTCOMES:
WOSI | 4 months
  Western Ontario Stability Index questionnaire is a tool designed for self-assessment of shoulder function for patients with instability problems.
  This questionnaire has 21 questions, each scored on a scale from 0 to 100, with 0 being the best score (no limitations related to the shoulder) and 100 representing the worst score.
  Overall, the questionnaire is scored as a percentage of the maximum score of 2100 points.
  There are subscale components reporting on: physical symptoms (questions 1 through 10; maximum score of 1000); sports/recreation/work (questions 11 through 14; maximum score 400); lifestyle (questions 15 through 18; maximum score 400); and emotion (questions 19-21; maximum score 300).
  Subscale scores are added to determine the total score out of a possible 2100 points, with 2100, or 100%, representing the worst possible score.
Pain level | 4 months
  Assessment of shoulder pain will be measured by the Numerical Rating scale of pain (NRS) with numbers from 0 - 10 ("no pain" to "worst pain imaginable"). The pain level will be measured at baseline as the intensity of pain right now, and at 16 weeks follow-up, and in addition, the worst, least and average pain level for the latest week will be measured one time weekly.
Checklist Individual Strength (CIS) | 4 months
  Assessment of fatigue by the Checklist Individual Strength (CIS), subscale fatigue will be performed at baseline and at 16-week follow up to report the change in level of fatigue. CIS Subscale fatigue consists of 8 items each scored on a 7-point Likert scale (scores ranging from 8 to 56) with high scores indicating high levels of fatigue
COOP/WONCA | 4 months
  To assess the change in functional health status from baseline to 16 weeks follow-up the COOP/WONCA questionnaire will be used. The questionnaire is a generic health status questionnaire for General Practice patients. The questionnaire consists of six single-item measures; physical fitness, feelings (mental well-being), daily activities, social activities, besides change in health and overall health. The categories chosen are scored from one (good functional status) to five (poor functional status)
Tampa Scale of Kinesiophobia (TSK-11) | 4 months
  Tampa scale of Kinesiophobia is used to measure impression of change in fear of movement from baseline to 16 weeks follow-up. It consists of an 11-item scale where each question is scored on a 4 point Likert scale, with 1 indicating, "strongly disagree" and 4 indicating, "strongly agree". The total scores range from 11-44, with higher scores representing increased fear of movement.
Global Perceived Effect (GPE) | 4 months
  To measure the patients self-rated impression of recovery at follow-up the GPE will be used. GPE measures self-rated impression of recovery since baseline assessment on a 7-point scale (1= worst ever; 2= much worse; 3= a little worse; 4= not changed; 5= a little improved; 6= much improved; and 7= best ever)
EQ-5D-5L Health status questionnaire | 4 months
  The EQ-5D-5L measures change in health related quality of life. It comprises five dimensions (mobility, Self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension is rated using a five-level ordinal scale from no problems to extreme problems. It results in a preference based index that range from states worse than death (<0), to 1 (full health), anchoring dead at 0. A score of one indicates that the participants perceived their health at the best possible state and a score below null that the participants perceived their health worse than death. In addition, the EQ-5D includes an EQ-VAS where own health "today" is rated on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
IPAQ short version | 4 months
  Physical Activity Questionnaire. To measure the weekly physical activity level the short version of the IPAQ will be used. The IPAQ collects information on time spent on physical activity (PA) at moderate and vigorous intensity and walking in 4 domains: work, transportation, housework/gardening, and leisure time. Questions are supplied with examples of common activities. In all domains, participants are asked to indicate the amount of time spent on PA in the past 7 days in relation to frequency (days) and duration (hours or minutes) of the activity.
Isometric shoulder strength | 4 months
  Maximum isometric voluntary contraction (MVC) in shoulder scaption, internal rotation and external rotation using a hand-held dynamometer.
Active and passive shoulder range of motion | 4 months
  Internal rotation and external rotation with shoulder in 90 degrees of abduction is measured using a HALO digital goniometer.
Shoulder proprioception | 4 months
  Shoulder proprioception is measured in shoulder flexion angles using af HALO digital goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Liaghat, MSc, Principal Investigator — University of Southern Denmark; Birgit Juul-Kristensen, PhD, Study Director — University of Southern Denmark; Søren T Skou, PhD, Study Chair — University of Southern Denmark, Næstved-Slagelse-Ringsted Hospitals; Karen Søgaard, PhD, Study Chair — University of Southern Denmark; Jens Søndergaard, MD, PhD, Study Chair — University of Southern Denmark; Uffe Jørgensen, MD, Study Chair — Odense University Hospital, University of Southern Denmark
Locations (3):
- Denmark (3):
  - GP´s and physiotherapists, Middelfart, Egion of Southern Denmark
  - GP´s and physiotherapists, Esbjerg, Region Syddanmark
  - GP´s and physiotherapists, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liaghat B, Skou ST, Jorgensen U, Sondergaard J, Sogaard K, Juul-Kristensen B. Heavy shoulder strengthening exercise in people with hypermobility spectrum disorder (HSD) and long-lasting shoulder symptoms: a feasibility study. Pilot Feasibility Stud. 2020 Jul 10;6:97. doi: 10.1186/s40814-020-00632-y. eCollection 2020. PMID 32670599
- See also: Manuscript open access — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-020-00632-y